CLINICAL TRIAL: NCT05332470
Title: A Real-world Study of Lamivudine and Dotiravir Sodium Tablets in the Treatment-naïve HIV-1 Infected Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUMCH record ZS-3419D
Record Dates: First submitted 2022-04-10; First posted 2022-04-18 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: HIV-1-infection
Keywords: Lamivudine and Dotiravir Sodium Tablets; Dovato
MeSH Terms: interventions — Lamivudine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Lamivudine and Dotiravir Sodium Tablets — 3TC (300 mg p.o. q 24 h) plus DTG (50 mg p.o. q 24 h)
  Other Names: Dovato

SUMMARY:
Actual update to the US Department of Health and Human Services treatment guidelines for HIV-1 infection and European AIDS Clinical Society guidelines indicate Dovato(Dolutegravir/lamivudine) as an initial treatment in HIV-naÏve patients. However there is no real- life data. The investigators' results in real life have encouraged us to conduct a multicenter cohort study in patients who have already started their first antiretroviral therapy with DTG (dolutegravir) + 3TC(lamivudine ), to verify efficacy and tolerance in real life. The investigators' hypothesis is that the data will be similar to those reported in clinical trials.

DETAILED DESCRIPTION:
Since 1996, HAART(Highly Active Antiretroviral Therapy) based on 3DR(3-drug regimens ) in PLHIV(people living with HIV) has decreased mortality and today, PLHIV have a life expectancy close to that of the general population. In the last decade new drugs have improved tolerance and posology of these treatment. However PLHIV needs to continue the treatment and will likely remain on antiviral therapy for many years. In the recent period, active research is being sought with the aim of improving the dosage and reducing the amount of drugs necessary to maintain efficacy, to avoid the possible cumulative effects of long-term ART (antiretroviral therapy). 2DRs(Two-drug regimens) have been investigated as a means for reducing the number of ARVs(antiretroviral agents) taken by individuals who need lifelong ART. Dovato has been evaluated in two phase III studies (GEMINI-1 and GEMINI-2) in treatment-naive adults achieving non inferiority according to the US FDA (Food and Drug Administration) Snapshot algorithm. These data led to the approval of the fixed-dose combination of dolutegravir/lamivudine as a once-daily, single-tablet 2DR by the FDA and the European Medicines Agency. Actual update to the US Department of Health and Human Services treatment guidelines for HIV-1 infection and European AIDS Clinical Society guidelines indicate Dovato as an initial treatment in HIV-naÏve patients. However there is no real- life data. The investigators' aim is to provide information related to effectiveness and tolerability/safety in naïve patients when used in routine clinical practice. It has been already published results from the phase III study in pretreatment adult patients.

The investigators' results in real life have encouraged us to conduct a multicenter cohort study in patients who have already started their first antiretroviral therapy with DTG (dolutegravir) + 3TC(lamivudine ), to verify efficacy and tolerance in real life. The investigators' hypothesis is that the data will be similar to those reported in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and sign the written informed consent ;
2. Over 18 years old;
3. Western Blot test confirmed HIV positive, and did not take any antiretroviral therapy;
4. HIV viral load ≥1000 copies/ml ;
5. Uncomplicated hepatitis B virus infection: HBsAg (-) ;
6. Estimated glomerular filtration rate (GFR) > 30ml/min (calculated by CKD - EPI);
7. No serious liver function damage (Child C ) ;
8. Be able to carry out antiviral treatment and regular follow-up according to the plan.

Exclusion Criteria:

1. Previously used ART or used PreP or PEP ;
2. Have a history of mental or nervous system diseases or suicidal tendencies;
3. Severe cardiovascular and respiratory system diseases, liver and kidney function damage, coagulation dysfunction, thrombocytopenia, circulatory system diseases, etc.;
4. There are indications of glucocorticoid application during application or follow-up period;
5. Radiotherapy, chemotherapy, cell therapy or therapeutic vaccine, immunomodulatory therapy, etc. are required within 28 days before the start of the study or during the study period;
6. Participate in other drug trials;
7. Those who are pregnant, breastfeeding or planning to become pregnant within one year;
8. Poor compliance, unable to follow up on schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the treatment-naïve HIV-1 infected patients
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of individuals with HIV-1 RNA <50 copies/ml at 24 weeks | 24 weeks
  Proportion of individuals with HIV-1 RNA <50 copies/ml at 24 weeks

SECONDARY OUTCOMES:
Proportion of individuals with HIV-1 RNA <50 copies/ml at 48 weeks | 48 weeks
  Proportion of individuals with HIV-1 RNA <50 copies/ml at 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: WEI Lyu, Principal Investigator — Department of Infectious Diseases, PekingUMCH

IPD SHARING:
Plan to Share IPD: No